CLINICAL TRIAL: NCT04765358
Title: Virtual Diabetes Specialty Clinic: A Study Evaluating Remote Initiation of Continuous Glucose Monitoring
Acronym: VDiSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VDiSC
Record Dates: First submitted 2021-01-15; First posted 2021-02-21 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Other): All participants were provided with a commercially available CGM system. Training and data collection for the study was completed remotely. After initial CGM training (initiation of unblinded CGM use or initial training with virtual clinic) was completed, participants were followed by the virtual clinic team for approximately six months. Psychosocial screening questionnaires were administered at enrollment and during follow up. The virtual clinical team member followed up with the study participant if there was an elevated score on the psychosocial screening questionnaires. After the initial six months of follow up, participants who decided to continue to use CGM were asked to extend follow up and complete questionnaires, submit HbA1c samples, and share data. During the extended follow up phase, participants were able to contact the virtual clinic with questions or to request assistance as needed.
  Interventions: Other: Virtual Clinic

INTERVENTIONS:
Other: Virtual Clinic — CGM, Clinical Care Support and Behavioral Health Support

SUMMARY:
The objective of this study was to evaluate a virtual diabetes clinic model, for adults with either type 1 diabetes or type 2 diabetes, that supports integration of CGM into diabetes self-management and use of decision support technology.

DETAILED DESCRIPTION:
Although demand for endocrinology care continues to grow, access to specialized care may be impacted by geographic isolation and a shortage in the number of endocrinologists in the United States. CGM use has been endorsed for individuals with T1D by the American Diabetes Association, the American Association of Clinical Endocrinologists, the Endocrine Society, and the International Society for Pediatric and Adolescent Diabetes. Despite these recommendations and the compelling evidence of the benefits of CGM, many individuals with T1D or insulin-using T2D have not incorporated CGM into their diabetes management.

The study was designed to assess feasibility and efficacy of establishing a virtual diabetes clinic with a focus on introduction and training related to use of CGM technology and ongoing CGM use to minimize such rate-limiting factors as geography, cost and access to specialty care. The virtual diabetes clinic model included a comprehensive care team with support for diabetes technology such as CGM and decision support to align with current recommendations in diabetes care. The virtual diabetes clinic model also included mental health screening and support services, particularly for diabetes-related issues.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old
2. Diagnosis of type 1 diabetes or type 2 diabetes and using insulin therapy (at least 3 injections of insulin per day or insulin pump that is compatible with Tidepool software); Multiple daily injection (MDI) users must be willing to use a device provided by the study that records the injection dosages and/or enter insulin dosing information through an app
3. See a healthcare provider at least once a year
4. Resident of United States and plan to reside in the U.S. for the duration of the study (This requirement is due to virtual clinic license requirements and U.S. use restrictions for some study software and devices. Not all U.S. states may be eligible for inclusion due to virtual clinic license status.)
5. Use either an Android or iOS smartphone that is compatible with app requirements that are needed for the study
6. Access to a compatible computer with internet
7. Understand written and spoken English
8. Willing and able to follow the study procedures as instructed

Exclusion Criteria:

1. Current use of a closed loop system where an insulin pump and CGM share information and insulin dose is automatically adjusted based on glucose reading
2. Current CGM use where Time in Range is ≥60.0% or Time <54% is ≤1.0%.
3. Current use of any off-label glucose-lowering medications for diabetes type (Example: T1D use of non-insulin, anti-diabetic medications including SGLT2 inhibitors). Use of such medications during the study will also be prohibited.
4. Females who are pregnant, intending to become pregnant, or breastfeeding during the study
5. Current renal dialysis or plan to begin renal dialysis during the study
6. Active cancer treatment
7. Extreme visual or hearing impairment that would impair ability to use real-time CGM
8. Known adhesive allergy/prior skin reaction or skin reaction identified during the blinded CGM use phase that would preclude continued CGM use
9. Participation in a different diabetes management study during the study
10. Planned relocation to a state other than current state of residence during the study if virtual clinic is not licensed in the new state. Individuals working routinely in a state other than current state of residence in the next six months are also ineligible if the virtual clinic is not licensed in that state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grazia Aleppo, MD, Study Chair — Northwestern University Feinberg School of Medicine; Robin L Gal, MSPH, Principal Investigator — Jaeb Center for Health Research
Locations (1):
- Jaeb Center for Health Research, Tampa, Florida, United States

REFERENCES:
- [Derived] Hood KK, Bergenstal RM, Cushman T, Gal RL, Raghinaru D, Kruger D, Johnson ML, McArthur T, Bradshaw A, Olson BA, Oser SM, Oser TK, Kollman C, Weinstock RS, Beck RW, Aleppo G. Patient-Reported Outcomes Improve with a Virtual Diabetes Care Model that Includes Continuous Glucose Monitoring. Telemed J E Health. 2025 Jan;31(1):75-84. doi: 10.1089/tmj.2024.0093. Epub 2024 Aug 21. PMID 39166322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 235
Completed | 234
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 187
  African American | 20
  Asian | 8
  American Indian-Alaskan Native | 1
  Other | 11
  Do not wish to answer | 7
Hemoglobin A1c [Mean (Standard Deviation); unit: mmol/mol] | 63 (17.5)
Time Spent with Glucose 70-<180 mg/dL [Mean (Standard Deviation); unit: percentage of 24 hour period] — Percentage of 24 hour period with blood glucose in target range of 70-180 mg/dL
  percentage of 24 hour period | 49 (25)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C (HbA1c)
Description: Percentage of red blood cells with glucose coated hemoglobin
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | All Participants
Number analyzed (Participants) | 226
mmol/mol | 54 (10.9)

2. Secondary Outcome: Time Spent With Glucose 70-180 mg/dL
Description: Percentage of 24 hour period with blood glucose in target range of 70-180 mg/dL
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: percentage of 24 hour period
Arm/Group | All Participants
Number analyzed (Participants) | 234
percentage of 24 hour period | 63 (18)

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/234
Serious Adverse Events (participants affected / at risk) | 16/234
Other Adverse Events (participants affected / at risk) | 22/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=234)
Severe hypoglycemia (Endocrine disorders) | 16 (17)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=234)
Hospitalization (General disorders) | 22 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/58/NCT04765358/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT04765358/SAP_004.pdf
  • Informed Consent Form (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT04765358/ICF_003.pdf